CLINICAL TRIAL: NCT04231487
Title: Using Wearable and Mobile Data to Diagnose and Monitor Movement Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jean-Francois Daneault, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Other Study IDs: Pro2018002015
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Essential Tremor; Parkinson Disease; Huntington Disease; Dystonia, Primary; Spinocerebellar Ataxias; Movement Disorders
MeSH Terms: conditions — Essential Tremor; Parkinson Disease; Huntington Disease; Dystonic Disorders; Spinocerebellar Ataxias; Movement Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Essential tremor: This is not an intervention study.
  Specific to group: a) Diagnosis of ET, b) stable dose of medication for 30 days
- Parkinson's Disease: This is not an intervention study.
  Specific to group: a) Diagnosis of PD, b) stable dose of medication for 30 days
- Huntington's Disease: This is not an intervention study.
  Specific to group: a) Diagnosis of HD, b) stable dose of medication for 30 days
- Primary Focal Dystonia: This is not an intervention study.
  Specific to group: a) Diagnosis of PFD, b) stable dose of medication for 30 days
- Spinocerebellar Ataxia: This is not an intervention study. Specific to group: a) Diagnosis of SCA, b) stable dose of medication for 30 days
- Functional Movement Disorder: This is not an intervention study. Specific to group: a) Diagnosis of FMD, b) stable dose of medication for 30 days
- Healthy Controls: This is not an intervention study.
  People with Healthy Controls

SUMMARY:
The purpose of the research is to better understand the motor behavior of individuals in health and disease. The specific purpose of this project is to identify if we can utilize a smartphone to diagnose different movement disorders and monitor their symptoms.

A. Objectives

1. Estimate symptom severity of Essential tremor (ET), Parkinson's disease (PD), Huntington's disease (HD), Primary focal dystonia (PFD), spinocerebellar ataxia (SCA), and Functional movement disorders (FMD) using a smartphone-based application
2. Differentiate individuals with the different movement disorders from healthy controls based on features from the smartphone data
3. Differentiate individuals with a specific movement disorder from people with other movement disorders based on features from the smartphone data

B. Hypotheses / Research Question(s) We hypothesize that we can estimate the severity of symptoms using a smartphone application and that, using those estimates, we can differentiate individuals with movement disorders from healthy controls and from people with other movement disorders.

DETAILED DESCRIPTION:
Movement disorders are a group of neurological conditions that alter human movements. They lead to functional impairments, diminished quality of life, and significant societal, economic, and familial burden. Due to the increase in population and longer life expectancy [1], more and more people will have to live with movement disorders. However, access to movement disorder specialists is already limited and will get worse [2]. Therefore, there is an urgent need to develop tools to aid non-specialist medical professionals identify and manage the symptoms (both motor and non-motor) of those disorders such that specialist can focus on more severe and complex cases. While there are several conditions that can be classified as movement disorders, the current proposal will focus on six disorders that have overlapping symptoms and could prove difficult to differentiate for non-specialists and/or clinicians that do not readily have access to genetic testing or imaging facilities: Essential tremor (ET), Parkinson's disease (PD), Huntington's disease (HD), primary focal dystonia (PFD), spinocerebellar ataxia (SCA), and functional movement disorders (FMD). While trained movement disorder specialists may correctly identify each of these disorders and provide optimal treatment, general practitioners and clinicians living in rural areas that do not have access to the most up-to-date diagnostic tools, such as neuroimaging and genetic testing, may face difficulty when treating those patients due to symptom variability and overlap in symptom presentation between different disorders; leading to sub-optimal treatment outcomes. As such, the development of simple, accurate, and inexpensive tools to help guide their clinical decisions is warranted. The ubiquity of mobile technology and wearable sensors may enable the development of such a tool. In recent years, our group and others have used mobile phones and wearable technology to assess symptoms in a multitude of disorders. This highlights the feasibility of our proposed system for the assessment and monitoring of symptom severity in individuals with movement disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* At least 18 years of age
* Ambulatory
* English speaking
* Specific to group 1: a) Diagnosis of ET, b) stable dose of medication for 30 days
* Specific to group 3: a) Diagnosis of PD, b) stable dose of medication for 30 days
* Specific to group 4: a) Diagnosis of HD, b) stable dose of medication for 30 days
* Specific to group 5: a) Diagnosis of PFD, b) stable dose of medication for 30 days
* Specific to group 6: a) Diagnosis of SCA, b) stable dose of medication for 30 days
* Specific to group 7: a) Diagnosis of FMD, b) stable dose of medication for 30 days

Exclusion Criteria:

* Serious untreated psychiatric illness that could impact the data collection
* Inability to understand task or protocol due to cognitive problems
* Other neurological condition that could affect the performance of motor tasks
* Musculoskeletal condition that could affect the performance of motor tasks
* Uncorrected vision impairment
* Specific to groups 1, 3, 4, 5, 6, and 7: Expected change in medication within the next 8 weeks

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - People with movement Disorders,
  We will recruit 7 parallel groups: 1) ET patients; 2) Healthy controls; 3) PD patients; 4) HD patients; 5) PFD patients; 6) SCA patients; and 7) FMD patients
  - Healthy Controls.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
UPDRS-III (Unified Parkinson's Disease Rating Scale) | Will occur right after the consent received from patients during the first lab visit.
  1. Speech (rating 0-4 were 0 is normal and 4 is Unintelligible), similarly following activities are recorded with a scale of (0-4)
  2. Facial Expression
  3. Tremor at Rest (head, upper and lower extremities)
  4. Action or Postural Tremor of Hands
  5. Rigidity (Judged on passive movement of major joints with patient relaxed in sitting position. Cogwheeling to be ignored.)
  6. Finger Taps (Patient taps thumb with index finger in rapid succession.)
  7. Hand Movements (Patient opens and closes hands in rapid succession)
  8. Rapid Alternating Movements of Hands (Pronation-supination movements of hands, vertically and horizontally, with as large an amplitude as possible, both hands simultaneously.)
  9. Leg Agility (Patient taps heel on the ground in rapid succession picking up entire leg. Amplitude should be at least 3 inches.)
  10. Arising from Chair
  11. Posture
  12. Gait
  13. Postural Stability
  14. Body Bradykinesia and Hypokinesia
TETRAS-performance (The Essential Tremor Rating Assessment Scale) | Will occur right after the consent received from patients during the first lab visit.
  Head Face Tongue Voice Upper limb Lower limb Spirals Handwriting Dot approximation Standing
Motor UHDRS for HD (Unified Huntington's Disease Rating Scale: Reliability and Consistency) | Will occur right after the consent received from patients during the first lab visit.
  OCULAR PURSUIT (horizontal and vertical) SACCADE INITIATION (horizontal and vertical) SACCADE VELOCITY (horizontal and vertical) DYSARTHRIA TONGUE PROTRUSION MAXIMAL DYSTONIA (trunk and extremities) MAXIMAL CHOREA (face, mouth, trunk and RETROPULSION PULL TEST FINGER TAPS (right and left) PRONATE/SUPINATE-HANDS (right and left) LURIA RIGIDITY-ARMS (right and left) BRADY KINESIA-BODY GAIT TANDEM WALKING
(UDRS) Unified Dystonia Rating Scale | Will occur right after the consent received from patients during the first lab visit.
  Eyes and upper face Lower face Jaw and tongue Larynx Neck Shoulder and proximal arm (right and left) Distal arm and hand including elbow Pelvis and proximal leg (right and left) Distal leg and foot including knee Trunk
(BARS) Brief Ataxia Rating Scale | Will occur right after the consent received from patients during the first lab visit.
  To develop a brief ataxia rating scale (BARS) for use by movement disorder specialists and general neurologists. BARS is valid, reliable, and sufficiently fast and accurate for clinical purposes.
(s-FMDRS) Simplified Functional Movement Disorders Rating Scale | Will occur right after the consent received from patients during the first lab visit.
  The Psychogenic Movement Disorders Rating Scale (PMDRS) has potential as a useful objective assessment in clinical research

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University, Newark, New Jersey, United States